CLINICAL TRIAL: NCT04829981
Title: The Health and Behavioural Impact of Implementing SAFEWATER Systems for Drinking Water Disinfection Within Rural Communities in Colombia and Mexico; Colombia.
Brief Title: SAFEWATER Health & Behaviour Impact Field Trials; Colombia
Acronym: SAFEWATER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Ulster (Other)
Collaborators: Fundación Cántaro Azul, A.C. (NGO), Mexico (Unknown); Centro de Ciencia y Tecnologia de Antioquia (CTA) (NGO), Colombia (Unknown); Universidad de Medellin, Colombia (Unknown); University of Sao Paulo (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: REC/18/0064 (C)
Record Dates: First submitted 2021-01-20; First posted 2021-04-02 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Water-Related Diseases
Keywords: Water, sanitation and hygiene (WASH); Water disinfection; Behaviour change; Stunting; Gut integrity; Malnutrition; Clean water technology; Diarrhoea; Child growth
MeSH Terms: conditions — Waterborne Diseases; Growth Disorders; Malnutrition; Diarrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention community (Experimental): Two communities in rural Colombia
  Interventions: Device: SAFEWATER systems for drinking water disinfection; Behavioral: Behaviour change interventions
- Control community (No Intervention): One community in rural Colombia

INTERVENTIONS:
Device: SAFEWATER systems for drinking water disinfection — A domestic water purification technology, consisting of a raw water storage tank, a pump, a filtration unit (2 cartridge filters), a UVC disinfection unit (UV lamp), a storage tank for drinking water (treated and safe water), and a distribution network inside the house for drinking water.
  Arms: Intervention community
Behavioral: Behaviour change interventions — Targeting behaviors around the use of the technology and water more generally. Behavioral interventions will be data-driven (i.e., dependent on the problems that arise) but are likely to include household and community-level activities.
  Arms: Intervention community

SUMMARY:
At least 1.8 billion people globally use a source of drinking water that is faecally contaminated and thus likely to lead to diarrheal illness: nearly 1,000 children die each day due to water and sanitation-related diarrhoeal diseases. Diseases related to the consumption of contaminated drinking-water place a major burden on human health. In 2017, 785 million people still lacked access to an improved drinking water source, and these are mostly the poor and marginalised. Almost a quarter of those people rely on surface water that is untreated and over 90% live in rural areas. Many people are forced to rely on sources that are microbiologically unsafe, leading to a higher risk of contracting waterborne diseases, including typhoid, hepatitis A and E, polio and cholera. The objectives of the SAFEWATER project is to develop technologies to provide clean water to economically deprived communities in rural Colombia and Mexico. These water technologies will be tested under real conditions with the cooperation of the rural communities.

The SAFEWATER field trials aims to evaluate the health and behaviour impacts of implementing SAFEWATER water treatment technologies for drinking water disinfection, with a behavioral change intervention, within rural communities in Colombia and Mexico

The project has three specific objectives:

1. Assess water quality improvement at household level
2. Assess behaviors and test behavioral interventions'
3. Assess child growth and related health outcomes

Three communities in Colombia and one community in Mexico were recruited to take part in the study. Communities were selected based on factors such as current availability of clean water, accessibility, safety, community size and current activities within the communities.

Pilot and feasibility studies were carried out prior to commencing field trials, thus the design of the trials vary across countries.

Mexico field trial: The trial in Mexico will use a stepped-wedge design, randomized at household level over a 12-month period (6-12 steps dependent on adherence and feasibility). All households (max n200) willing to be involved will be recruited (separate clinicaltrials.gov registration).

Colombia field trial: the trial in Colombia will use a non-randomized parallel design (2:1; intervention:control). A maximum of 84 households (54:30; intervention:control) will be recruited to take part, with families with young children (<12 years) prioritized.

Outcomes for both countries will include 1) water quality, 2) water-related behaviour (e.g. frequency of system use, uses of treated / raw water), and 3) health, e.g. diarrhoea prevalence, growth (height/weight), school attendance, water insecurity status, gut integrity.

Impact: The development and deployment of the SAFEWATER technology has the potential to impact on clean drinking water access for participating communities in Mexico and Colombia, and subsequently on the health and wellbeing of those individuals involved. Additionally if successful, the work will also provide an evidence based model for the provision of improved access to clean drinking water for rural communities in developing regions more widely.

ELIGIBILITY:
Inclusion Criteria:

* Communities in rural communities without access to clean water systems
* Households where the head of the household fully understands the study information provided and is willing to provide consent.
* Households where it is feasible to install the SAFEWATER system

Priority Criteria:

1. Having at least one child of 12 years or under in the household
2. Having previously worked with Universidad de Medellin or CTA (criteria #2 will only be implemented if households meeting #1 is exhausted)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Water quality | Change over 12 months
  Microbial load
Use of safe water | Change over 12 months
  Frequency
Child (12 years and under) growth | Change over 12 months
  Change in BMI percentile to identify stunting, wasting and underweight

SECONDARY OUTCOMES:
Water quality | Change over 12 months
  Turbidity (measured using a turbidimeter (NTU units)
Use of safe water | Change over 12 months
  Practices for drinking, hygiene and cooking i.e. what the water is used for and how
Use of the system | Change over 12 months
  Frequency; intervention group only
Use of the system | Change over 12 months
  Practices; intervention group only i.e. what the water is used for and how
Untreated water usage | Change over 12 months
  Frequency
Untreated water usage | Change over 12 months
  Practices for drinking, hygiene and cooking i.e. what the water is used for and how
Water storage practices | Change over 12 months
  Frequency
Water storage practices | Change over 12 months
  Method
Handwashing with soap | Change over 12 months
  Frequency
Sharing of safe water to external households | Change over 12 months
  Intervention group only. Frequency and volume of water shared with external households
Fetching water | Change over 12 months
  Frequency
Diarrhoea prevalence | Change over 12 months
  Bristol Stool Chart (Type 1(hard) - 7(soft)
School attendance | Change over 12 months
  Absence (days)
Household water insecurity status | Change over 12 months
  The Household Water Insecurity Experiences (HWISE) Scale (scores 0-36 (higher scores indicate greater insecurity))
Gut integrity | Change over 12 months
  Fingerprick test for iron levels in a sub-group of children as a proxy marker of improved gut integrity.
Maintenance to SAFEWATER system | Change over 12 months
  Frequency (intervention group only)
Maintenance to SAFEWATER system | Change over 12 months
  Nature of maintenance; intervention group only
Satisfaction of SAFEWATER system | Change over 12 months
  Level of satisfaction for system and water provided, including taste, colour & temperature and odour (1(satisfied) - 3(unsatisfied)) + reasons (qualitative)
Making unplanned changes to the system | Change over 12 months
  Making changes for functional or aesthetical reasons which could potentially interfere with the functioning of the system (list of changes / household) - intervention group only
Study retention | Change over 12 months
  Percentage completed appointments

CONTACTS AND LOCATIONS:
Locations (3):
- Colombia (2):
  - Universidad de Medellin, Medellín, Antioquia
  - Centro de Ciencia y Tecnologia de Antioquia (CTA),, Medellín
- Fundación Cántaro Azul, A.C, San Cristóbal de las Casas, Chipas, Mexico

IPD SHARING:
Plan to Share IPD: Yes